CLINICAL TRIAL: NCT06330974
Title: Allergy, Asthma, and Atopic Eczema in Finland - A Nationwide Study on Prevalence, Comorbidities, Treatment and Economic Burden
Brief Title: Allergy, Asthma, and Atopic Eczema in Finland
Acronym: FinnATOPY
Status: Not yet recruiting | Type: Observational
Sponsor: Tampere University (Other)
Collaborators: Professor Lauri Lehtimäki (Unknown); Professor Mika Mäkelä (Unknown); Professor Sanna Toppila-Salmi (Unknown); Professor Ilkka Junttila (Unknown)
Responsible Party: Principal Investigator, Peter Csonka, MD, PhD, Associate professor of pediatrics, Tampere University
Other Study IDs: FinnATOPY
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Asthma; Asthma in Children; Allergy; Rhinitis, Allergic; Atopic Dermatitis; Allergen Immunotherapy
MeSH Terms: conditions — Asthma; Hypersensitivity; Rhinitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The summary is available at --> https://www.finnatopy.fi/summary

DETAILED DESCRIPTION:
Aims and objectives ---> https://www.finnatopy.fi/aims-and-objectives Methods ---> https://www.finnatopy.fi/methods

ELIGIBILITY:
Inclusion/Exclusion Criteria ---> https://www.finnatopy.fi/methods

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: https://www.finnatopy.fi/methods
Sampling Method: Non-Probability Sample
Enrollment: 2000000 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Epidemiology of atopic diseases and allergic sensitization profiles in Finland | 7 years
  Incidence and prevalence of asthma, specific IgE sensitization, atopic dermatitis, allergic rhinitis
Burden of atopic diseases (allergies, asthma, and atopic eczema) as well as comorbidities in Finland | 7 years
  Morbidity, sick leaves, medication use, costs and expences
Evaluate and improve the current use of diagnostic tests for atopic diseases | 7 years
  Diagnostic practices, tests for allergic sensitization, lung function tests, and other laboratory measures.
Use and effectiveness of allergen immunotherapy in real world setting | 7 years
  Real world evidence data using specific cohorts
Direct and indirect costs related to atopic diseases and comorbidities | 7 years
  All costs, including sick leaves, absenteeism, laboratory costs, other diagnisteic tests, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Péter Csonka, Principal Investigator — Tampere University
Locations (1):
- Tampere University, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided